CLINICAL TRIAL: NCT02150603
Title: Assessment of Patterns of Patient-reported Outcomes in Adults With Congenital Heart Disease - International Study
Brief Title: Patient-Reported Outcomes in Adults With Congenital Heart Disease
Acronym: APPROACH-IS
Status: Completed | Type: Observational
Sponsor: Philip Moons (Other)
Responsible Party: Sponsor-Investigator, Philip Moons, prof. dr. Philip Moons, Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Other Study IDs: ML9231
Record Dates: First submitted 2014-05-21; First posted 2014-05-30 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Heart Defects, Congenital
Keywords: Heart defects, congenital; Patient-reported outcomes; Health status; Factors, psychosocial; Health behavior; Quality of life; Sense of coherence; Illness perceptions; Depression; Anxiety
MeSH Terms: conditions — Heart Defects, Congenital; Health Behavior; Depression; Anxiety Disorders

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults with congenital heart disease

SUMMARY:
The purpose of this study is to examine the differences in perceived health, psychosocial functioning, behavioral outcomes and quality of life of adults with congenital heart disease who are living in different areas of the world, and how these differences can be understood (e.g., differences in sense of coherence or illness perceptions).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with congenital heart disease, defined as: a gross structural abnormality of the heart or intra-thoracic great vessels that is actually or potentially of functional significance (including mild, moderate, and severe heart defects)
* 18 years of age or older
* Diagnosed under the age of ten, i.e. before adolescence
* Continuing follow-up at an adult congenital heart disease center or included in a national/regional registry
* Physical, cognitive, and language abilities to complete self-report questionnaires

Exclusion Criteria:

* Prior heart transplantation
* Isolated pulmonary hypertension
* Syndromes affecting cognitive abilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with congenital heart disease who are in continuing follow-up at an adult congenital heart disease center or included in a national/regional registry.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2013-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Patient-reported health status (EuroQol-5D) | Baseline
Patient-reported psychosocial functioning (Hospital Anxiety and Depression Scale) | Baseline
Patient-reported behavioral outcomes (Health Behavior Scale - Congenital Heart Disease) | Baseline
Patient-reported quality of life (Linear Analog Scale Quality of Life;Satisfaction with Life Scale) | Baseline

SECONDARY OUTCOMES:
Patient-reported sense of coherence (Sense of Coherence scale 13 items) | Baseline
Patient-reported illness perceptions (Brief Illness Perception Questionnaire) | Baseline
Patient-reported socio-demographic variables (e.g. age, educational level) | Baseline
Medical variables by chart review (e.g. cardiac surgeries, frequency of follow-up) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Philip Moons, PhD, Study Director — KU Leuven; Koen Luyckx, PhD, Study Director — KU Leuven; Adrienne Kovacs, PhD, Study Director — Peter Munk Cardiac Centre, University Health Network
Locations (24):
- United States (6):
  - Stanford Hospital & Clinics, Stanford, California
  - Washington University and Barnes Jewish Heart & Vascular Center, St Louis, Missouri
  - Children's Hospital & Medical Center, Omaha, Nebraska
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
- Hospital de Niños, Córdoba, Argentina
- Private practice, Melbourne, Australia
- University Hospitals Leuven, Leuven, Belgium
- Canada (3):
  - Northern Alberta Adult Congenital Heart Clinic, Edmonton
  - Montreal Heart Institute, Montreal
  - Peter Munk Cardiac Center, Toronto
- Hôpital Luis Pradel, Lyon, France
- Frontier Lifeline Hospital, Chennai, India
- IRCCS Policlinico San Donato Hospital, Milan, Italy
- Chiba Cardiovascular Center, Chiba, Japan
- Mater Dei Hospital, Msida, Malta
- Amsterdam Medical Center, Amsterdam, Netherlands
- Oslo University Hospital, Oslo, Norway
- Sweden (3):
  - Sahlgrenska University Hospital/ Östra, Gothenburg
  - Karolinska Institute, Stockholm
  - University Hospital of Umeå, Umeå
- University Hospital Bern, Bern, Switzerland
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Kovacs AH, Luyckx K, Thomet C, Budts W, Enomoto J, Sluman MA, Lu CW, Jackson JL, Khairy P, Cook SC, Chidambarathanu S, Alday L, Estensen ME, Dellborg M, Berghammer M, Johansson B, Mackie AS, Menahem S, Caruana M, Veldtman G, Soufi A, Jameson SM, Callus E, Kutty S, Oechslin E, Van Bulck L, Moons P; APPROACH-IS Consortium, International Society for Adult Congenital Heart Disease. Anxiety and Depression in Adults With Congenital Heart Disease. J Am Coll Cardiol. 2024 Jan 23;83(3):430-441. doi: 10.1016/j.jacc.2023.10.043. PMID 38233017
- [Derived] Moons P, Luyckx K, Thomet C, Budts W, Enomoto J, Sluman MA, Yang HL, Jackson JL, Khairy P, Cook SC, Chidambarathanu S, Alday L, Oechslin E, Eriksen K, Dellborg M, Berghammer M, Johansson B, Mackie AS, Menahem S, Caruana M, Veldtman G, Soufi A, Fernandes SM, White K, Callus E, Kutty S, Kovacs AH; APPROACH-IS consortium. Patient-reported outcomes in the aging population of adults with congenital heart disease: results from APPROACH-IS. Eur J Cardiovasc Nurs. 2023 May 25;22(4):339-344. doi: 10.1093/eurjcn/zvac057. PMID 35901014
- [Derived] Lu CW, Wang JK, Yang HL, Kovacs AH, Luyckx K, Ruperti-Repilado FJ, Van De Bruaene A, Enomoto J, Sluman MA, Jackson JL, Khairy P, Cook SC, Chidambarathanu S, Alday L, Oechslin E, Eriksen K, Dellborg M, Berghammer M, Johansson B, Mackie AS, Menahem S, Caruana M, Veldtman G, Soufi A, Fernandes SM, White K, Callus E, Kutty S, Apers S, Moons P; APPROACH-IS consortium, the International Society for Adult Congenital Heart Disease (ISACHD) *. Heart Failure and Patient-Reported Outcomes in Adults With Congenital Heart Disease from 15 Countries. J Am Heart Assoc. 2022 May 3;11(9):e024993. doi: 10.1161/JAHA.121.024993. Epub 2022 Apr 26. PMID 35470715
- [Derived] Fox KR, Hardy RY, Moons P, Kovacs AH, Luyckx K, Apers S, Cook SC, Veldtman G, Fernandes SM, White K, Kutty S, Jackson JL; APPROACH-IS Consortium and the International Society for Adult Congenital Heart Disease (ISACHD). Smoking among adult congenital heart disease survivors in the United States: Prevalence and relationship with illness perceptions. J Behav Med. 2021 Dec;44(6):772-783. doi: 10.1007/s10865-021-00239-5. Epub 2021 Jun 29. PMID 34185220
- [Derived] Moons P, Luyckx K, Thomet C, Budts W, Enomoto J, Sluman MA, Lu CW, Jackson JL, Khairy P, Cook SC, Chidambarathanu S, Alday L, Eriksen K, Dellborg M, Berghammer M, Johansson B, Mackie AS, Menahem S, Caruana M, Veldtman G, Soufi A, Fernandes SM, White K, Callus E, Kutty S, Ombelet F, Apers S, Kovacs AH; APPROACH-IS Consortium and the International Society for Adult Congenital Heart Disease (ISACHD). Physical Functioning, Mental Health, and Quality of Life in Different Congenital Heart Defects: Comparative Analysis in 3538 Patients From 15 Countries. Can J Cardiol. 2021 Feb;37(2):215-223. doi: 10.1016/j.cjca.2020.03.044. Epub 2020 Apr 6. PMID 32739453
- [Derived] Moons P, Apers S, Kovacs AH, Thomet C, Budts W, Enomoto J, Sluman MA, Wang JK, Jackson JL, Khairy P, Cook SC, Chidambarathanu S, Alday L, Oechslin E, Eriksen K, Dellborg M, Berghammer M, Johansson B, Mackie AS, Menahem S, Caruana M, Veldtman G, Soufi A, Fernandes SM, White K, Callus E, Kutty S, Luyckx K; APPROACH-IS consortium and the International Society for Adult Congenital Heart Disease (ISACHD). Sense of coherence in adults with congenital heart disease in 15 countries: Patient characteristics, cultural dimensions and quality of life. Eur J Cardiovasc Nurs. 2021 Feb 11;20(1):48-55. doi: 10.1177/1474515120930496. PMID 32524857
- [Derived] Van Bulck L, Goossens E, Luyckx K, Apers S, Oechslin E, Thomet C, Budts W, Enomoto J, Sluman MA, Lu CW, Jackson JL, Khairy P, Cook SC, Chidambarathanu S, Alday L, Eriksen K, Dellborg M, Berghammer M, Johansson B, Mackie AS, Menahem S, Caruana M, Veldtman G, Soufi A, Fernandes SM, White K, Callus E, Kutty S, Moons P; APPROACH-IS consortium and the International Society for Adult Congenital Heart Disease (ISACHD). Healthcare system inputs and patient-reported outcomes: a study in adults with congenital heart defect from 15 countries. BMC Health Serv Res. 2020 Jun 3;20(1):496. doi: 10.1186/s12913-020-05361-9. PMID 32493367
- [Derived] Holbein CE, Veldtman GR, Moons P, Kovacs AH, Luyckx K, Apers S, Chidambarathanu S, Soufi A, Eriksen K, Jackson JL, Enomoto J, Fernandes SM, Johansson B, Alday L, Dellborg M, Berghammer M, Menahem S, Caruana M, Kutty S, Mackie AS, Thomet C, Budts W, White K, Sluman MA, Callus E, Cook SC, Khairy P, Cedars A; APPROACH-IS consortium and the International Society for Adult Congenital Heart Disease (ISACHD). Perceived Health Mediates Effects of Physical Activity on Quality of Life in Patients With a Fontan Circulation. Am J Cardiol. 2019 Jul 1;124(1):144-150. doi: 10.1016/j.amjcard.2019.03.039. Epub 2019 Apr 10. PMID 31030969
- [Derived] Apers S, Kovacs AH, Luyckx K, Alday L, Berghammer M, Budts W, Callus E, Caruana M, Chidambarathanu S, Cook SC, Dellborg M, Enomoto J, Eriksen K, Fernandes SM, Jackson JL, Johansson B, Khairy P, Kutty S, Menahem S, Rempel G, Sluman MA, Soufi A, Thomet C, Veldtman G, Wang JK, White K, Moons P; APPROACH-IS consortium; International Society for Adult Congenital Heart Disease (ISACHD). Assessment of Patterns of Patient-Reported Outcomes in Adults with Congenital Heart disease - International Study (APPROACH-IS): rationale, design, and methods. Int J Cardiol. 2015 Jan 20;179:334-42. doi: 10.1016/j.ijcard.2014.11.084. Epub 2014 Nov 8. PMID 25464481
- See also: Related Info — http://approach-is.net/